CLINICAL TRIAL: NCT06720753
Title: Examining Mechanisms of Change in Adolescent Self-Inflicted Injury
Brief Title: Real-time Examination of Skills and Coping Use in Teen's Everyday Lives
Acronym: RESCUE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Erin Kaufman, Assistant Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: K23MH135225 (NIH)
Record Dates: First submitted 2024-11-22; First posted 2024-12-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Self Injurious Behavior; Suicide
Keywords: Self Injurious Behavior; Dialectical Behavior Therapy; Therapy mechanisms; Suicide; Adolescents; Families; fMRI; Psychophysiological measures
MeSH Terms: conditions — Self-Injurious Behavior; Suicide

STUDY DESIGN:
Masking Description: Research assistants performing behavioral coding will be masked to participant condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opposite action (Experimental): Participants will be randomly assigned to this arm either first or second. All participants complete both arms.
  Interventions: Behavioral: Opposite to emotion action
- GIVE (Experimental): Participants will be randomly assigned to this arm either first or second. All participants complete both arms.
  Interventions: Behavioral: GIVE

INTERVENTIONS:
Behavioral: Opposite to emotion action — Participants will be taught the opposite action skill from Dialectical Behavior Therapy
  Arms: Opposite action
Behavioral: GIVE — Participants will be taught the GIVE skill from Dialectical Behavior Therapy
  Arms: GIVE

SUMMARY:
The goal of this clinical trial is to compare two core intervention skills among adolescents with a history of engaging in at least 3 lifetime incidents of self-inflicted injury (SII), at least one of which was a suicide attempt of at least moderate lethality and moderate intent to die. The main questions it aims to answer are:

Whether and when youth use skills in daily life, how quickly skill use declines after teaching, and whether exposure to life stress influences skill learning and retention.

The Investigators also want to know whether brain-related, family-related, and physiology-related factors influence skills practice and any associated changes in self-harm/suicide risk and emotion dysregulation.

Participants will complete surveys 5 times a day on their phones at baseline, and following each skill learning session. All participants will learn and practice the two skills with a parent while discussing topics they often argue about. During these discussions, participants will be hooked up to psychophysiological equipment to measure their cardiovascular functioning and their palm sweat. Participants' discussions will be coded for skill use and also for indices of family functioning. Approximately half of the participants will undergo two sets of fMRI scans to assess potential neural underpinnings of skill use.

DETAILED DESCRIPTION:
Suicide marks an extreme along a continuum of self-inflicted injury (SII) and is a leading cause of death among adolescents. Although psychologists have evidence-supported interventions for youth SII, the biosocial mechanisms supporting change are underexplored. Lack of innovation in this area has led to statis, rather than decline, in population-level suicide rates. The field also lacks vital data on: if/when adolescents apply therapeutic skills in daily life, the neural and physiological factors influencing skill uptake, and whether such skills are effective in reducing SII and related risk and vulnerability factors.

When identifying key intervention targets, theoretical and empirical work implicate emotion dysregulation and interpersonal stressors in SII etiology and maintenance. Adaptive emotion regulation strategies and strong social ties each reduce the likelihood of suicidal ideation and SII among otherwise vulnerable individuals, and improvements in emotion regulation are associated with SII cessation. Yet, the specific skills and mechanisms promoting self-regulatory improvements are not well understood.

This study is designed to rigorously examine two competing SII intervention mechanisms. The research plan and aims are devoted to identifying youth who may benefit from a brief skill-building intervention and biosocial mechanisms supporting skill acquisition. The investigator use a within-subjects design to directly compare the effects of teaching an intra- vs. interpersonal skill from Dialectical Behavior Therapy (DBT; a widely-used intervention for SII). Adolescents with a history of repeated SII (n = 100) will participate in 4 laboratory visits with a primary caregiver. At Visit 1, participants will complete interviews and questionnaires assessing psychiatric diagnoses, SII, and life stress, and 50 will complete two functional MRI paradigms to tap neural processes underlying perspective taking and empathy, and approach/avoidance. Adolescents will then complete a 2-week EMA protocol (EMA1, Training Aim 2) to measure daily affect, perceived stressors, SII, and suicidal thoughts, pre-intervention. At Visit 2, dyads will be randomly assigned to learn and practice GIVE (interpersonal skills training) or opposite-to-emotion action (OA; intrapersonal skill). The investigator will assess behavioral, affective, and physiological regulatory processes (respiratory sinus arrythmia [RSA]) during two conflict discussions: (1) pre- skills training, and (2) post-training, while dyads use their assigned skill. This laboratory assessment will be followed by a second EMA period (EMA2) to assess skill use and EMA1 variables. Post EMA2, dyads will return for Visit 3 to repeat fMRI assessment before undergoing training in the alternate skill ⎯ followed by another 2-week EMA protocol (EMA3). Finally, participants will complete a remote follow-up visit 6 months post-EMA3, where the investigator will reassess SII, symptom severity, and life stressors as well as barriers to skill use. This study will assess and integrate multimodal responses to core intervention mechanisms in a high-risk sample.

Aim 1: Examine within-person mechanistic (brain, RSA) changes as a function of skills training in the laboratory (Training Aim 1).

H1a: Participants will show less RSA withdrawal during skill-practice relative to a pre-training conflict task. H1b: Such intervention changes will translate to increased left ventro-lateral prefrontal cortex engagement during an fMRI paradigm tapping OA; and increased medial pre-frontal cortex engagement during a task tapping perspective taking and empathy (corresponding to GIVE).

H1c: Compared with the OA condition, GIVE training will result in less RSA withdrawal during skills practice.

H1d: The investigator will test whether skill practice effects (H1a, b) are moderated by recent life stressors (Training Aim 3) and expect severe stressors in the 6 months preceding study participation will be associated with less improvement during skills practice across outcome measures.

Aim 2: Examine the effects of skills training on outcomes relevant to suicide risk in daily life.

H2a: Changes observed post-skills training in the GIVE and OA conditions will extend into social and affective improvements in participants' daily lives as reported via EMA - especially in the context of momentary skills use.

H2b: Further, the investigator hypothesize that skill use during laboratory visits and EMA will predict subsequent reductions in life stressors that are dependent on adolescent characteristics and/or behaviors.

Aim 3: Examine persistence/decay effects of skill in daily life following initial skill exposure and a "booster" call.

H3a: Skill use will be most frequent immediately following training and decline over time. H3b: A brief booster call 1 week post-skill exposure will predict increases in EMA reported skill use. The investigator will examine potential moderation effects to determine who may benefit from repeated skill exposure.

H3c: Youth skill use over the EMA period will predict changes in stressor severity experienced over 6-month followup. Specifically, GIVE use will predict less severe dependent stress.

ELIGIBILITY:
Inclusion Criteria:

* 3+ incidents of self-inflicted injury (SII). At least one SII episode must score a minimum of "3" on lethality (moderate; e.g., overdose on 11-50 pills; deep cuts anywhere but neck) and "4" on intent (somewhat serious [about dying]) - even if aborted or interrupted. Adolescents with 3+ SIIs may also enroll if they have been hospitalized for suicide preparatory behavior.
* English language proficiency
* Access to a smart phone
* Parent/caregiver/legal guardian to participate with the adolescent

Exclusion Criteria:

* Moderate to severe developmental or intellectual disability, psychosis, or a schizophrenia spectrum diagnosis.
* Those taking medications with well-documented effects on psychophysiological responding.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Rates of skill use in daily life as assessed via ecological momentary assessment mobile surveys | Frequency of skills use reported over the course of two 10-day EMA periods immediately post skills training (EMAs are 5 x per day)
  The investigators will assess the rate of self-reported skills use across post-skill training EMA periods to understand retention, generalization, and potential decay effects. We will also examine whether rates increase following a brief booster call intended to reiterate the skill to youth participants.
Self-injurious urges, behaviors, and suicidal ideation as reported on ecological momentary assessment items | Changes will be assessed from pre-intervention baseline (Visit 1 and a ten day baseline EMA period [EMA1]) across EMA 2 and 3, and 6-month follow-up (post-intervention).
  Change in self-reported rates and intensity of self-inflicted injury urges/behavior and suicidal ideation will be assessed from pre- to post-skills training. We will compare data from baseline interviews/surveys/EMA1 to post-skills training time points (EMA2 and EMA 3) and 6-month follow-up (assessed with the L-SASII). Frequency of self-reported skill use in daily life will be used as a key predictor variable.
Emotion regulation/dysregulation changes as assessed on the difficulties in emotion regulation scale- short form (DERS-SF) | Patterns and changes in emotion regulation/dysregulation indices will be assessed from Visit 1 through 6-month follow-up (approximately 8 months).
  The investigators will be examining change in self-reported emotion regulation/dysregulation from the pre-intervention discussion task to post-skills training via the difficulties in emotion regulation scale short form (DERS-SF). The answers are assessed using a 5-point Likert scale, from 1 (almost never) to 5 (almost always). It is possible to obtain the score of each of 6 subscales, and the total score of the DERS-SF (18-90), with higher values indicating greater difficulties in emotion regulation.
Neural patterns and changes from pre- to post-skills training on fMRI tasks (Opposite action paradigm and EmpaTom-Y) | Visit 1 and post-intervention scan at Visit 3 (taken approximately 5-6 weeks apart.
  Participants will learn skills in the laboratory environment and implement them in daily life. The investigators will observe change in neural activation in response to skill-targeted probes of empathy and perspective taking and opposite action from pre- to post-training (Visit 1 to Visit 3). Specifically, the investigators expect intervention changes will translate to (1) increased left ventro-lateral prefrontal cortex engagement during an fMRI paradigm tapping opposite action; and (2) increased medial pre-frontal cortex engagement during a task tapping perspective taking and empathy (EmpaTom-Y; corresponding to GIVE).
Impact of life stress (assessed with the Life Events and Difficulties Schedule; LEDS-II) on skill learning and retention as reported on ecological momentary assessment items | A baseline life stress assessment will be completed at Visit 1 (Life Events and Difficulties Schedule; LEDS-II). Skill learning and retention will be assessed via ecological momentary assessment items assessing skill use for approximately 6 weeks.
  The investigators will assess associations between experiences of life stress at baseline (assessed via the LEDS-II interview) and subsequent rates of skill use in daily life (EMA2 and EMA3).
Barriers to skill use as self-reported on ecological momentary assessment | Across approximately 2 months
  Participant reported barriers to skill use will be assessed via ecological momentary assessment items. This information will aid us in better optimizing how these skills are taught.

SECONDARY OUTCOMES:
Impact of skills use on life stress as assessed by the Life Events and Difficulties Schedule (LEDS-II) | Approximately 8 months
  The investigators hypothesize that skill use during laboratory visits and in daily life (assessed via ecological momentary assessment; EMA) will predict subsequent reductions in life stressors the that are dependent on adolescent characteristics and/or behaviors (assessed by comparing LEDS-II results from baseline to 6-month follow-up).
Changes in family functioning from pre-intervention to post-intervention discussion tasks as assessed via The System for Coding Interactions and Family Functioning (SCIFF) | Across approximately 4-5 weeks
  All family discussion tasks will be coded with the SCIFF to examine changes from pre- to post-intervention training.
Examine changes in emotion regulation/dysregulation from pre- to post-intervention discussion tasks via respiratory sinus arrhythmia (RSA) | Across approximately 1 month
  RSA will be assessed as a physiological index of emotion regulation across all discussion tasks (both pre- and post-intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Erin Kaufman, Ph.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
We will post descriptions of study methods (including Dialectical Behavior Therapy Skills videos) and procedures to our Open Science Framework (OSF) page. All de-identified data and code relevant to the project will be uploaded to OSF upon submission to encourage replications and extensions of our work. In addition to the data for neuroimaging and RDoC domains, demographic and clinical information will be included.
  Data collected for exploratory aims will be uploaded upon completion of publication and all relevant reports and publications will be made available per the open access policy of NIH.
Supporting Information: Study Protocol, SAP
Time Frame: All materials will be shared following analysis and publication of main study questions.
Access Criteria: All de-identified data and code relevant to the project will be uploaded to OSF